CLINICAL TRIAL: NCT06433726
Title: A Phase Ⅰ, Multi-center, Open-label, Dose-escalation, Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Anti-tumor Activity of BY101921 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Phase l Study of By101921, an Oral PARP7 Inhibitor, in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Baiyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1921-I-01
Record Dates: First submitted 2024-05-13; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BY101921 (Experimental): Dose Escalation: Multiple doses of BY101921 for oral administration
  Interventions: Drug: BY101921 tablets

INTERVENTIONS:
Drug: BY101921 tablets — An oral PARP7 Inhibitor

SUMMARY:
BY101921 is a novel small molecule, being developed as a PARP7 inhibitor which acts on the PARP7 catalytic subunit, for the treatment of solid tumors. PARP7 is a member of the monoPARP family and involved in various biological processes such as gene expression, protein degradation, and cellular stress response. The results of non-clinical studies showed BY101921 was a potent inhibitor of PARP7 and had good selectivity.

The primary objective is to assess the safety and tolerability and MTD of BY101921 in patients with refractory or metastatic solid tumors. This study will also evaluate pharmacokinetic (PK) profile, preliminary anti-tumor activity, major metabolites and biomarkers in patients with refractory or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years and ≤75 years of age.
2. patients histologically or cytologically diagnosed advanced malignant solid tumors who have failed, cannot tolerate, or refuse prior standard treatment regimens. At least 1 measurable lesion per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
3. Have a projected life expectancy of at least 3 months.
4. Eastern Cooperative Oncology Group Performance Status 0 or 1.
5. Adequate organ and bone marrow function. Laboratory tests that meet the following criteria within 7 days prior to the first dose of study treatment (without blood transfusion, erythropoietin, recombinant human thrombopoietin or colony stimulating factor therapy, renal replacement therapy, etc., within 28 days prior to the screening examination):

   Routine blood test:

   Absolute neutrophil count (ANC) ≥ 1.5×109/L Platelets count (PLT) ≥ 100×109/L Hemoglobin (Hb) ≥ 90 g/L

   Hepatic function:

   Total bilirubin (TBIL) ≤ 1.5×ULN Aspartate aminotransferase (AST) ≤ 2.5×ULN Alanine aminotransferase (ALT) ≤ 2.5×ULN ALT and AST ≤ 5×ULN and TBIL ≤ 3×ULN for patients with primary liver cancer, liver metastases, or Gilbert 's syndrome.

   Renal function:

   Creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula).

   Coagulation function:

   International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN
6. Females and males of childbearing potential must agree to use appropriate methods of contraception (hormonal/barrier method or abstinence) during the study and for 3 months after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to administration.
7. Understand and be willing to sign written informed consent and be able to follow the study protocol for treatment, visits, and other study procedures.

Exclusion Criteria:

1. Previously treated with PARP-7 inhibitors.
2. Treated with a potent CYP3A4 inhibitor or inducer within 2 weeks prior to the first dose of study treatment.
3. Previous any treatment with of the following:

   1. Systemic chemotherapy, other antitumor agents (including endocrine therapy, macromolecular targeted therapy, immunotherapy, or biotherapy) within 4 weeks or 5 half-lives prior to the first dose of study treatment, or who need to continue receiving these agents during the study period;
   2. Small molecule targeted therapy within 2 weeks or 5 half-lives prior to the first dose of study treatment;
   3. Anti-tumor traditional Chinese medicine or proprietary Chinese medicine preparations prior to the first dose of study treatment;
   4. Nitrosourea or mitomycin C within 6 weeks prior to the first dose of study treatment;
   5. Palliative radiation therapy within 2 weeks prior to the first dose of study treatment;
   6. Investigational drug within 4 weeks prior to the first dose of study treatment; g Radical radiation therapy within 4 weeks prior to the first dose of study treatment.
4. Major surgical intervention (excluding needle biopsy) within 28 days before study drug administration, surgical wound has not fully healed or surgery is scheduled during the study period.
5. Brain metastasis (except asymptomatic, stable for more than 4 weeks prior to the first dose and not requiring steroid therapy for at least 4 weeks prior to the first dose, no imaging findings of marked edema around the tumor lesion), presence of meningeal metastasis or brainstem metastasis, or presence of spinal cord compression.
6. History of other malignancy within the past 5 years, except skin basal cell carcinoma, skin squamous cell carcinoma, cervical carcinoma in situ, or other carcinomas in situ which have undergone curative treatment and have had no recurrence within 5 years after treatment.
7. Toxicities from prior antitumor therapy that have not recovered to CTCAE version 5.0 Grade 1 or less, except CTCAE (V5.0) Grade 2 peripheral neurotoxicity and alopecia of any grade.
8. Difficult-to-control pleural effusion, ascites, or pericardial effusion.etc, requiring repeated drainage and considered unsuitable for study enrollment by the investigator.
9. Serious or uncontrolled diseases as assessed by the investigator, including but not limited to:

   Severe or uncontrolled diabetes, poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg under standardized antihypertensive regimens), epilepsy, chronic obstructive pulmonary disease, interstitial pneumonia, pulmonary interstitial fibrosis, Parkinson 's disease, active bleeding, uncontrolled infection.

   Cognitive dysfunction, history of psychiatric disorders, other uncontrolled concomitant diseases, alcohol dependence, hormone dependence, or drug abuse.

   History of immunodeficiency, including HIV antibody positive, other acquired or congenital immunodeficiency disease, or history of organ transplantation.

   HBsAg or HBcAb positive, and peripheral blood HBV DNA titer test ≥ 200 IU/mL or ≥ 1000 copies/mL or above the upper limit of normal value at the study site; HCV antibody test positive, and HCV RNA test above the upper limit of normal value at the study site; treponema pallidum-specific antibody positive.

   Clinically serious gastrointestinal dysfunction that may compromise drug intake, transport, or absorption. For example, inability to take oral medication, uncontrollable nausea or vomiting, history of massive gastrointestinal resection, history of gastrointestinal ulcer and gastrointestinal bleeding within 6 months prior to the first dose, untreated recurrent diarrhea, untreated stomach disease requiring long-term use of PPI acid suppressants, Crohn 's disease, ulcerative colitis, etc.
10. Cardiac dysfunction, including any of the following:

    Myocardial infarction in past 6 months, heart failure classified as Class II/III/IV according to the New York Heart Association (NYHA) Functional Classification, unstable angina pectoris, and unstable arrhythmia.

    Left ventricular ejection fraction LVEF < 50% shown by echocardiography. QT interval corrected using Fridericia 's formula: QTcF > 470 msec (females), QTcF > 450 msec (males).
11. Pregnant (positive pregnancy test prior to dosing) or lactating.
12. History of serious hypersensitivity (e.g., anaphylactic shock) or hypersensitivity to excipients or other ingredients associated with the study drug.
13. Cannot follow the protocol to "avoid ingesting grapefruit , pomegranate, orange or green lemon (juice/sauce made from these fruits as well) within 7 days before study drug administration and throughout the BY101921 treatment period".
14. Other factors considered unsuitable for study enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BY101921 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  Grade and frequency of adverse events and serious adverse events
To assess the maximum tolerated dose (MTD) | through study completion (an average of 1.5 years)
  Incidence of Dose limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
To assess preliminary antitumor activity of BY101921 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  ORR
To assess pharmacokinetics (PK) parameters of BY101921 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  AUC
To assess pharmacokinetics (PK) parameters of BY101921 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  Cmax
To assess pharmacokinetics (PK) parameters of BY101921 in patients with advanced solid tumors | through study completion (an average of 1.5 years)
  T1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Shandong First Medical University / Shandong Cancer Research Institute / Shandong Cancer Hospital, Jinan, Shandong, China